CLINICAL TRIAL: NCT01136447
Title: Success Rate of Infra-clavicular Blocks: Comparison of Ultrasound Versus Neurostimulation Guided Catheter Placement
Brief Title: Continuous Infraclavicular Blocks: Neurostimulation Versus Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Shalini Dhir, DR., London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-06-101; 12208 (Other: REB)
Record Dates: First submitted 2009-04-20; First posted 2010-06-03 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Disorder of Upper Extremity
Keywords: Brachial plexus; Ultrasound
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurostimulation (Placebo Comparator): Block catheter will be introduced using neurostimulation
  Interventions: Procedure: Ultrasound
- Ultrasound (Active Comparator): Block catheter will be introduced using ultrasound
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Block catheter will be introduced using ultraosound

SUMMARY:
The purpose of this study is to determine whether ultrasound guidance or nerve stimulation is the best option for placing continuous peripheral nerve block catheters for upper limb surgery.

DETAILED DESCRIPTION:
In a multidisciplinary, observer blinded, prospective, single center, randomized study, success rate of US guided versus neurostimulation guided catheter placement for continuous infraclavicular block in patients scheduled for upper limb surgery will be studied. Block effectiveness, time taken, discharge from recovery, postoperative pain and disability and patient acceptance will be studied in 210 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 yrs
* Weight 40-100 kg
* Either sex
* Height >150 cm
* American Society of Anesthesiologists physical status 1-3
* Scheduled for hand or elbow surgery under regional anesthesia

Exclusion Criteria:

* Inability to give informed consent
* Refusal of treatment randomization
* Language barrier
* Allergy to any medications being used in the study protocol
* Ongoing major medical or psychiatric problems
* Chronic pain or narcotic use/abuse
* Peripheral neuropathy or major neurological problems
* Scarring in area of blockade
* Inability to co-operate with post-operative evaluation
* Major coagulopathy
* Pregnancy and breast feeding
* Patients requiring anesthesia of other surgical sites
* Obese patients (i.e. BMI >40)
* Postoperatively, patients will be excluded if they have had additional operative procedures requiring a change in the usual protocol of care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Neurostimulation versus ultrasound guided infraclavicular catheter placement | 14 days
  Comparision of block success with neurostimulation and ultrasound guided placed infraclavicular catheters

SECONDARY OUTCOMES:
Time taken for complete nerve block | 14 days
  Procedure time for both techniques

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, MD, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada